CLINICAL TRIAL: NCT00593593
Title: A Pharmacovigilance Study to Evaluate Safety of AVODART (Dutasteride) Administration 0,5 mg Once Daily, for 52 Weeks, in Subjects With Benign Prostate Hyperplasia
Brief Title: Pharmacovigilance Study To Evaluate Safety Of AVODART In Subjects With Benign Prostate Hyperplasia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: 104244; Avodart-pv/GR
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostate hyperplasia; Dutasteride; pharmacovigilance
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study has 4 phases: screening phase (visit 1), treatment phase (visit 2 - 6 mths after treatment initiation), and end of treatment phase (visit 3 - end of year 1). Only in the case a serious adverse event (SAE) arises, will there be a follow up phase (visit 4).

ELIGIBILITY:
Inclusion Criteria:

* Subject should fulfil criteria for the subscription of AVODART as these are mentioned in the SPC
* Subject should be diagnosed with benign prostate hyperplasia
* Subject's prostate volume should be equal or greater than 30 cm3

Exclusion Criteria:

* Known hypersensitivity to any of the AVODART compounds
* Suffers from a serious illness which either is not properly controlled or as per investigator´s judgment could interfere with the subject´s compliance into the trial
* Receives treatment with enzyme inhibitors CYP3A4 and CYP3A5.
* History of severe liver failure

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline